CLINICAL TRIAL: NCT00258362
Title: A Phase II Trial of Induction Carboplatin and Docetaxel Followed by Radiotherapy Then Consolidation Chemotherapy With Carboplatin and Docetaxel in Stage III, IV and Recurrent Endometrial Cancer
Brief Title: Carboplatin, Docetaxel, and Radiation Therapy in Treating Patients With Stage III/IV, or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS021; UMN-WCC-38 (Other: Women's Cancer Center, University of Minnesota); 13062 (Other: Sanofi-Aventis Pharmaceuticals)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2010-11-11 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Docetaxel; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Endometrial Cancer (Experimental): Patients with advanced or current endometrial cancer receiving treatment with induction docetaxel/carboplatin, radiation (Weekly, 5 days/week over 6-7 weeks, tailored 4500 cGy) and followed by 3 courses of consolidation docetaxel (75 mg/m^2 on Day 1 of each course) /carboplatin (Dose = Area-under-the-curve 6 on Day 1 every 3 weeks for 3 cycles).
  Interventions: Drug: carboplatin; Drug: docetaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — Dose = Area-under-the-curve 6 on Day 1 every 3 weeks for 3 cycles.
  Other Names: Gemzar(R)
Drug: docetaxel — 75 mg/m^2 on Day 1 of each course
  Other Names: Taxotere(R)
Radiation: radiation therapy — Weekly, 5 days/week over 6-7 weeks (tailored 4500 cGy)
  Other Names: radiation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving carboplatin and docetaxel followed by radiation therapy works in treating patients with stage III, stage IV, or recurrent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with stage III or IV or recurrent endometrial cancer treated with induction chemotherapy comprising carboplatin and docetaxel followed by radiotherapy and consolidation chemotherapy comprising carboplatin and docetaxel.

Secondary

* Determine the toxic effects of this regimen in these patients.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: Patients receive docetaxel intravenous (IV) over 1 hour and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 courses. After hematologic recovery from chemotherapy, patients receive radiotherapy 5 days a week for up to 7 weeks. Beginning 3-4 weeks later, patients receive another 3 courses of docetaxel and carboplatin.

After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial cancer
* Advanced or recurrent disease

  * Stage IIIB or IIIC disease

    * Stage IIIA disease allowed provided there is serosal involvement or direct extension or metastasis to the adnexa
    * No stage IIIA confirmed by only positive peritoneal washings
  * Stage IVA or IVB disease
* Failed local therapy or considered incurable with local therapy
* Measurable or evaluable disease

  * Not required for newly diagnosed stage III or IV disease with no remaining disease after surgery
* Performance status Gynecology Oncology Group (GOG) 0-1
* Life expectancy at least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Meets 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal
* Bilirubin normal
* No acute hepatitis
* Creatinine ≤ 1.5 mg/dL

Exclusion Criteria:

* Known hypersensitivity to docetaxel or polysorbate 80
* Severe infection
* Septicemia
* Pregnant or nursing
* Positive pregnancy test
* Fertile patients must use effective nonhormonal contraception during and for at least 3 months after study treatment
* Peripheral neuropathy ≥ grade 2
* Severe gastrointestinal bleeding requiring a blood transfusion or hospitalization
* Other malignancy within the past 5 years except nonmetastatic, nonmelanoma skin cancer or carcinoma in situ of the cervix
* Prior chemotherapy
* Prior radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A. Geller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 patients consented originally, but 1 patient withdrew consent before receiving any treatment.
Groups:
- Patients With Endometrial Cancer: Patients with advanced or recurrent endometrial cancer receiving treatment with induction docetaxel/carboplatin, radiation (4500 cGy) and followed by 3 courses of consolidation docetaxel/carboplatin.
Period: Overall Study
Arm/Group | Patients With Endometrial Cancer
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Endometrial Cancer: Patients with advanced or recurrent endometrial cancer receiving treatment with induction docetaxel/carboplatin, radiation (4500 cGy) and followed by 3 courses of consolidation docetaxel/carboplatin. This group excludes those patients with recurrent endometrial cancer.
Arm/Group | Patients With Endometrial Cancer
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 35
  Black | 1
  Hispanic | 2
  Other | 2
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 41
Histology [Number; unit: Participants] — Type or classification of cancer
  Participants
    Endometroid | 32
    Serous | 4
    Mucinous | 1
    Adenosquamous | 3
    Endometroid + Serous | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Estimated to be Progression-Free and Alive
Description: This estimate was determined by using a statistical method of analysis (Kaplan-Meier).
Time Frame: 1 Year, 2 Years, 3 Years
Population: Two patients with recurrent disease at study entry were excluded from this analysis.
Measure: Number; unit: Percentage of Patients
Groups:
- Patients With Endometrial Cancer: Patients with advanced endometrial cancer receiving treatment with induction docetaxel/carboplatin, radiation (4500 cGy) and followed by 3 courses of consolidation docetaxel/carboplatin.
Arm/Group | Patients With Endometrial Cancer
Number analyzed (Participants) | 39
Percentage of Patients
  1 Year | 86 [69.0 to 93.8]
  2 Years | 76 [56.8 to 87.1]
  3 Years | 68 [44.6 to 83.2]

2. Secondary Outcome: Percent of Patients Estimated to be Alive
Description: This estimate of overall survival was determined by using the statistical method (Kaplan-Meier) of analysis.
Time Frame: 1 Year, 2 Years, 3 Years
Population: All 41 patients were included in this analysis.
Measure: Number; unit: Percentage of Patients
Arm/Group | Patients With Endometrial Cancer
Number analyzed (Participants) | 41
Percentage of Patients
  1 Year | 94 [79.5 to 98.6]
  2 Years | 91 [74.2 to 97.0]
  3 Years | 80 [45.4 to 93.6]

ADVERSE EVENTS:
Time Frame: Serious, related adverse events and other adverse events were collected from day 1 of treatment to 30 days post-treatment. Deaths outside the collection timeframe were not reported.
Description: Other adverse events were collected only once per patient (incidence); the number of events for each adverse event were not collected (frequency).
Arm/Group | Patients With Endometrial Cancer
Serious Adverse Events (participants affected / at risk) | 8/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Endometrial Cancer (N=41)
Bladder Infection (Renal and urinary disorders) | 2 (2)
Blood Infection (Infections and infestations) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Lymphocele (Blood and lymphatic system disorders) | 1 (1)
Metastatic disease to lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Resulted in death
Nausea (Gastrointestinal disorders) | 1 (1)
Stricture/stenosis of ureter (Renal and urinary disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Endometrial Cancer (N=41)
Anemia (Blood and lymphatic system disorders) | 31
Anorexia (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 20
Dermatology (Skin and subcutaneous tissue disorders) | 22
Diarrhea (Gastrointestinal disorders) | 16
Endocrine (Endocrine disorders) | 7
Fatigue (General disorders) | 37
Fever (General disorders) | 3
Hemorrhage (Blood and lymphatic system disorders) | 3
Infection (Infections and infestations) | 5
Leukopenia (Blood and lymphatic system disorders) | 24
Lymphatics (Blood and lymphatic system disorders) | 4
Musculoskeletal soft tissue (Musculoskeletal and connective tissue disorders) | 6
Neuropathy (Nervous system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 21
Ocular, visual (Eye disorders) | 3
Pain (General disorders) | 19
Pulmonary, upper respiratory (Respiratory, thoracic and mediastinal disorders) | 6
Renal, genitourinary (Renal and urinary disorders) | 4
Sexual reproductive function (Reproductive system and breast disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Vomiting (Gastrointestinal disorders) | 7
Weight loss (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No